CLINICAL TRIAL: NCT02073188
Title: Comparative Efficacy of iBGStar Glucose Meter vs. Traditional Glucose Monitoring in Improving Metabolic Control and Compliance Towards Self-Monitoring of Blood Glucose in Young Patients With Type 1 Diabetes
Brief Title: Comparative Study of a Smartphone-Linked Self-Monitoring System Versus a Traditional One for Improving Metabolic Control and Compliance to Self-Monitoring of Blood Glucose
Acronym: iNew Trend
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: IBGST_L_05971
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- iBGStar (Group A) (Experimental): Self-Monitoring Blood Glucose will be managed with iBGStar and iBGStar Diabetes Manager Application (App) uploaded on iPhone for all duration of the study (6 months of experimental phase plus 6-months of observational phase). In the first 3 months, the patients in Group A will send their glycemic test values and notes by mail to the physician through Diabetes Manager App every 2 weeks. Afterwards until the visit V2 (six months), the patients in Group A will send their glycemic test values and notes by mail monthly. 9 reports in total.
  Interventions: Device: iBGStar
- Traditional Glucometer (Group B) (Active Comparator): Self-Monitoring Blood Glucose will be managed with a traditional glucometer according to usual care for the first 6 months (experimental phase). In the 6 months post-trial follow-up (observational phase), Self-Monitoring Blood Glucose will be managed with iBGStar and iBGStar Diabetes Manager App.
  Interventions: Device: Traditional Glucometer

INTERVENTIONS:
Device: iBGStar
  Arms: iBGStar (Group A)
Device: Traditional Glucometer
  Arms: Traditional Glucometer (Group B)

SUMMARY:
The purpose of this study is to demonstrate the superiority of iBGstar as a component of the diabetes treatment vs. traditional blood glucose self-monitoring system for improving glycemic control after 6 months in young patients with type 1 diabetes. The study is intended also to demonstrate the superiority of iBGStar as a component of the diabetes treatment vs. usual blood glucose self-monitoring system for improving the compliance to self monitoring of blood glucose after 6 months.

DETAILED DESCRIPTION:
The planned study duration will be 20 months (5 quarters) with screening/enrollment of 7 months, followed by 2-3 weeks of a qualification phase, a 6 month experimental phase, plus a 6 month follow-up in the post-trial observational phase.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 diabetes
* Males and females
* Age between 14-24 years
* Any diabetes duration
* Cared for by the diabetes center for at least 1 year
* HbA1c ≥ 8%
* Basal bolus treatment (any insulin)
* Poor compliance with Self-Monitoring of Blood Glucose (less than 30% of the recommended Blood Glucose measurements recorded in the glucose meter in the two previous weeks, i.e. <16 Blood Glucose measurements in the last two weeks)
* Written informed consent obtained from patient or legal representative (for minor)

Exclusion Criteria:

* Treatment with other insulin regimen or Continuous Subcutaneous Insulin Infusion
* Refusal or inability to give informed consent to participate in the study
* Patients with short life expectancy
* Patients with conditions/concomitant diseases making them non evaluable for the primary efficacy endpoint according to physician's judgment
* Requirement for concomitant treatment that could bias primary evaluation
* Patients with high likelihood of being unavailable for 6 and/or 12 months visits
* Subject is the investigator, sub-investigator, research assistant, pharmacist, study coordinator, other study site staff or relative of study site staff thus considered directly involved in the conduct of the study
* Current addition/abuse of alcohol or drugs
* Severe visual or dexterity impairment
* Patients with any mental condition rendering them unable to understand the nature, scope, and possible consequences of the study
* Pregnant or breast-feeding women
* Subjects unlikely or unable to comply with the Protocol requirements

Ages: 14 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 186 (Actual)
Dates: Start 2012-06; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Change in HbA1c levels from baseline | baseline to six months
Proportion of participants performing at least 30% of the recommended Self-Monitoring Blood Glucose tests after 6 months from randomization | at 6 months

SECONDARY OUTCOMES:
Percentage of participants with HbA1c ≤7.5% | at 6 months and 12 months
Average number of recommended Self-Monitoring Blood Glucose tests daily, weekly, and monthly | at 6 months and 12 months
Mean fasting plasma glucose (FPG) and postprandial glucose (PPG) | at 6 months and 12 months
Mean Glycemic Variability | at 6 months and 12 months
Average Insulin Dose | at 6 months and 12 months
Number of Daily Injections | at 6 months and 12 months
Number of Insulin Dose Adjustments | at 6 months and 12 months
Quality of life: Audit of Diabetes Dependent Quality of Life (ADDQOL) (young adults 18-24 years) | at 6 months and 12 months
Diabetes Quality of Life (DQOL-Y) (adolescents 14-17 years) | at 6 months and 12 months
Participants satisfaction with SMBG meter assessed by Visual Analog Scale (VAS) | at 6 months and 12 months
Number overall contacts between centers and participants | up to 12 months
Type of overall contacts between centers and participants | up to 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Sanofi -Aventis Administrative Office, Milan, Italy

REFERENCES:
- [Derived] Di Bartolo P, Nicolucci A, Cherubini V, Iafusco D, Scardapane M, Rossi MC. Young patients with type 1 diabetes poorly controlled and poorly compliant with self-monitoring of blood glucose: can technology help? Results of the i-NewTrend randomized clinical trial. Acta Diabetol. 2017 Apr;54(4):393-402. doi: 10.1007/s00592-017-0963-4. Epub 2017 Jan 30. PMID 28138788